CLINICAL TRIAL: NCT01956708
Title: Transfer of Cardioprotection During Remote Ischemic Conditioning
Brief Title: Transfer of Cardioprotection During RIPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Markus Kamler, Prof. Dr. med. Markus Kamler, University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: RIPC-13-5507-BO
Record Dates: First submitted 2013-09-27; First posted 2013-10-08 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: CABG

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote ischemic preconditioning (Active Comparator): Remote ischemic preconditioning (RIPC) protocol before coronary artery bypass surgery (CABG):
  after induction of anesthesia and before surgery: 3 cycles of 5 minutes left upper arm ischemia by inflation of a blood pressure cuff to 200mmHg and 5 minutes of reperfusion Anesthesia is with isoflurane (0.7-0.8% end-tidal) +sufentanil
  Interventions: Procedure: RIPC
- Placebo (Placebo Comparator): No Remote ischemic preconditioning (RIPC) protocol before coronary artery bypass surgery (CABG):
  after induction of anesthesia and before surgery: the cuff is left uninflated
  Interventions: Procedure: RIPC

INTERVENTIONS:
Procedure: RIPC — 3 cycles of 5 min left upper arm ischemia by inflation of a blood pressure cuff to 200 mmHg and 5 min reperfusion
  Other Names: RIPC: Remote ischemic preconditioning

SUMMARY:
Remote ischemic preconditioning (RIPC) with transient upper limb ischemia/reperfusion provides peri-operative myocardial protection, is safe and improves prognosis in patients undergoing elective CABG surgery.

The signal transfer from limb to heart is unknown. Thus, the aim of this study is to identify the pathways which transfer the cardioprotective signal from the ischemic/reperfused extremity to the heart in humans undergoing surgical coronary revascularization.

DETAILED DESCRIPTION:
The investigators will obtain arterial blood samples before skin incision and 1-72 h after the remote ischemic preconditioning protocol and analyze them biochemically. The investigators focus on those ligands that have been previously implicated in conditioning protocols at any organ. In addition, the investigators will use a bioassay system, consisting of a Langendorff-perfused isolated heart with coronary occlusion/reperfusion and infarct size by TTC staining as endpoint, and then expose this bioassay system to arterial plasma obtained after the remote ischemic preconditioning stimulus or placebo. This approach will allow us to further characterize any potential transfer signal candidate with a pharmacological antagonist approach.

The investigators will also obtain human atrial appendages after the remote ischemic preconditioning protocol or placebo and before patients were connected to the extracorporeal circulation. Contractile function of isolated trabeculae and vasomotor function of isolated arterial vessels will be analyzed in a bioassay system.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients > 18 years after written informed consent
* elective, isolated CABG surgery with and without valvuloplastic surgery
* two-stage cannulation, cardiopulmonary bypass
* antegrade Bretschneider cardioplegia
* mild hypothermia (32°C)
* preoperative standard medication (statins, betablocker, aspirin)
* standard anesthesia (see above)
* intraoperative standard protocol (full heparinization with ACT, aprotinin, protamin)
* postoperative standard protocol (500 mg aspirin after 2 h, low-dose heparin after 4 h)

Exclusion Criteria:

preoperative

* prior percutaneous coronary intervention (PCI) within 6 weeks
* any preoperative troponin T elevation
* renal insufficiency (creatinine >200 µmol/l)
* reoperation
* emergency surgery
* acute coronary syndrome (unstable angina, STEMI, NSTEMI) within 4 weeks
* dual anti-platelet therapy (clopidogrel+aspirin)

intraoperative

* harvesting of a. radialis
* coronary thrombendarterectomy
* complications (bypass-low flow/ -occlusion)
* antithrombotic therapy (intraoperative clopidogrel + aspirin)
* retrograde cardioplegia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2013-09; Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Myocardial protection | 72 h, postoperatively
  Cumulative postoperative troponin T release

SECONDARY OUTCOMES:
All-cause mortality | 30 days and 1 year after CABG surgery and after complete follow-up
  follow up done by studynurses
MACCE | 30 days and 1 year after CABG surgery after complete follow-up
  Major adverse cardiac and cerebrovascular events
renal function | 72 h, postoperatively
  Creatinine and eGFR
Cardioprotective factors released into circulating blood | before skin incision versus 1-72 h after RIPC
  Analysis of blood plasma
Myocardial function in vitro | after RIPC
  left ventricular pressure (lvp) and maximum left ventricular pressure (lvdp) in an isolated perfused rodent heart after blood plasma infusion

CONTACTS AND LOCATIONS:
Overall Officials: Markus Kamler, MD, Principal Investigator — Herzzentrum Essen - Huttrop gGmbH, Einrichtung des Universitätsklinikums Essen, Essen, Germany
Locations (1):
- Herzzentrum Essen - Huttrop gGmbH, Einrichtung des Universitätsklinikums Essen, Essen, Germany